CLINICAL TRIAL: NCT04849117
Title: Effect of Bilateral Transversus Thoracis Muscle Plane Block on Postoperative Morphine Consumption in Patients Undergoing Elective On-pump Coronary Artery Bypass Graft Surgery: a Retrospective Study.
Brief Title: Effect of Bilateral Transversus Thoracis Muscle Plane Block in Patients Undergoing Coronary Artery Bypass Graft Surgery.
Acronym: PARACABS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0582
Record Dates: First submitted 2021-03-23; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Pain Syndrome
Keywords: Cardiac Surgery; Coronary Artery Bypass Graft Surgery; Regional Anesthesia; Transversus Thoracis Muscle Plane Block; Enhanced Recovery After Surgery; Pain, evaluated by visual analog scale score.
MeSH Terms: conditions — Coronary Artery Disease; Somatoform Disorders; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic analgesia: Patients received only systemic analgesia : Acetaminophen, Ketoprofen, and Nefopam were administered systematically. Morphine was administered if necessary, according to our institutional pain management protocol.
- Bilateral TTMP block + systemic analgesia: Patients received the same protocol of systemic analgesia associated with a bilateral TTMP block performed during the first four hours after ICU admission, before tracheal tube removal.
  Interventions: Procedure: Ultrasound guided Bilateral Transversus Thoracis Muscle Plane block

INTERVENTIONS:
Procedure: Ultrasound guided Bilateral Transversus Thoracis Muscle Plane block — In the "TTMP block" group, an ultrasounded guided TTMP block was performed by an anesthesiologist, in ICU, before tracheal tube removal. Between the 4th et 5th rib, on each side, 40 ml of Ropivacaine 2 mg/ml, in association with Clonidine, was injected "single-shot" in the tranversus thoracis muscle plane. The targets of local anesthetic were the anterior branches of intercostal nerves from T2 to T6. Dexamethasone 8 mg was injected intravenously.
  Other Names: Transversus Thoracis Muscle Plane Block. Parasternal Block.
  Groups: Bilateral TTMP block + systemic analgesia

SUMMARY:
Coronary artery bypass graft surgery is the standard surgical treatment for coronary disease. However, there is no consensus on analgesic management in patients undergoing CABG.

The aim of the study is to evualuate efficacy of bilateral transversus thoracis muscle plane (TTMP) block combined with systemic analgesia, compared to systemic analgesia only, in patients undergoing elective on-pump CABG surgery.

Our main hypothesis is that a bilateral TTMP block performed after CABG surgery could reduce morphine consumption during the first 48 hours.

The investigators conducted an age, gender and type of surgery-matched retrospective cohort study in the Montpellier University Hospital (France).

ELIGIBILITY:
Inclusion criteria:

* To be over 18
* To be scheduled for CABG surgery in the center of the study during the study period.

Exclusion criteria:

* Chronic pain or opioid use before surgery
* Recent thoracic regional analgesia (< 1 month)
* Preoperative dementia or other neurologic or psychiatric disease incompatible with VAS pain scoring.
* Other technique of regional anesthesia (e.g. thoracic epidural)
* Opposition to data collection

Secondary exlusion criteria:

* Postoperative prolonged sedation in ICU (> 12 hours)
* Postoperative surgical complication requiring surgical revision during the first two days.
* Opposition to data collection expressed secondarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "TTMP Block" group : fifty consecutive patients who underwent elective on-pump coronary artery bypass graft ± valve surgery after October 2019, with a postoperative analgesic protocol including a bilateral TTMP block, associate with systemic analgesia.
  "Systemic Analgesia" group : age, gender and type of surgery-matched patients who underwent elective on-pump coronary artery bypass graft ± valve surgery before September 2019, with a postoperative analgesic protocol based on systemic analgesia only.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
cumulative morphine consumption | postoperative day 2
  cumulative morphine consumption during the first two days. cumulative morphine consumption on postoperative day 0, 1 and 2, including the morphine administered in intensive care unit, and on postoperative day 1 and 2.

SECONDARY OUTCOMES:
Postoperative pain assessed | postoperative day 0, 1 and 2
  Postoperative pain assessed by visual analog scale (VAS) scoring
Postoperative nausea and vomiting | hospital day 7
  Postoperative nausea and vomiting
Occurrence of prurit | postoperative day 7
  Occurrence of prurit
rate of Delirium | postoperative day 7
  rate of Delirium
rate of Constipation | postoperative day 7
  rate of Constipation
rate of Urinary retention | until postoperative day 7
  rate of Urinary retention
rate of Hypotension | until postoperative day 7
  rate of Hypotension
Pleural drain duration | day 20
  Pleural drain duration
Urinary catheter duration | day 20
  Urinary catheter duration
Duration of hospitalization in ICU | day 20
  Duration of hospitalization in ICU
In-hospital length of stay | day 20
  In-hospital length of stay
Occurrence of atrial fibrillation | until postoperative day 7
  Occurrence of atrial fibrillation
rate of Pneumonia | until postoperative day 7
  rate of Pneumonia
acute kidney injury | until postoperative day 7
  acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Sentenac, MD, PhD, Principal Investigator — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC